CLINICAL TRIAL: NCT04884204
Title: Systematic Symptom Identification With Disease Specific PROM to Assess Symptoms of Chronic GVHD in Outpatient Care in Patients Post HSCT - a Two Site Feasibility Study
Brief Title: Systematic Symptom Identification With Disease Specific PROM to Assess Symptoms of Chronic GVHD in Outpatient Care in Patients Post HSCT
Acronym: SIMPly-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Mary Jarden, Professor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Copenhagen, Rigshospitalet
Record Dates: First submitted 2021-04-30; First posted 2021-05-12 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: GVHD, Chronic; Hematological Malignancy
Keywords: Lee Symptom Scale; Symptom management; Patient reported outcome
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Symptom management with Lee Symptom Scale (Experimental): Participants will receive disease specific questionnaires electronically, cGVHD-PRO (Lee Symtpom Scale), one week prior to their scheduled visit in the outpatient clinic. The participants will be asked to answer the questionnaire from home without any involvement from clinicians. Afterwards the PRO data will be used during the scheduled clinical consultations as an instrument to discover symptoms on chronic GVHD and systematically to monitoring symptoms developing over time.
  Interventions: Behavioral: Lee Symptom Scala

INTERVENTIONS:
Behavioral: Lee Symptom Scala — Symptom identification and management with Lee Symptom Scale in follow up care

SUMMARY:
A two sited feasibility study to test the feasibility of systematic symptom identification with disease specific and clinically developed PROM (Lee Symptom Scale) longitudinally with a 12 month follow up in outpatient care in patients post HSCT to assess symptoms of chronic GVHD (n= 30).

DETAILED DESCRIPTION:
A prospective, non-randomized, feasibility study examining a systematic approach to symptom management using PROMs with 12 months of follow up in hematological outpatient clinic

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years old
* Approximately 3 months post HSCT (they will be included before HSCT, but the intervention will begin at 3 moths).
* Patients included needs to be able to manage a computer to receive and respond to collect PRO data.

Exclusion Criteria:

* Patients who do not understand, read and speak Danish and/or have cognitive/psychiatric disorders not compatible with inclusion in a clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Recruiment time frame: 12 months
  Number of participants included from eligible participants
Adherence to intervention | Intervention time frame: 12 months of follow up
  Number of visits completed out of planned visits during intervention

SECONDARY OUTCOMES:
Quality of life measured by the European Organization for Research and Treatment of Cancer - quality of life questionnaire C30 (EORTC-QLQ-C30) | 12 months; at baseline (0 months), 6 and 12 months
  Change in quality of life measured by the European Organization for Research and Treatment of Cancer - quality of life questionnaire C30
Depression and Anxiety measured with the Hospital Anxiety and Depression Scale | 12 months; at baseline (0 months), 6 and 12 months
  Change in symptoms of depression and anxiety measured by the Hospital Anxiety Depression Scale
MD Andersons Symptom Inventory (MDASI) | 12 months; at baseline (0 months), 6 and 12 months
  Change in symptom burden measured by the scale M.D. Andersons Symptom Inventory
HM-PRO questionaire developed by the 'Scientific Working Group for QoL and Symptoms,' within the European Hematology Association | 12 months; at baseline (0 months), 3, 6, 9 and 12 months
  Change in HM-PRO developed by The 'Scientific Working Group for QoL and Symptoms,' within the European Hematology Association

OTHER OUTCOMES:
Diagnose | At baseline
  Diagnose at baseline
Medication | At baseline
  Medication at baseline
Immunosuppresive drugs | 12 months of follow up from date of transplantation
  Immunosuppresive drugs the participants receive after transplantation (within the study period)
Hospitalization | 12 months of follow up from date of transplantation
  Periods with hospitalizations within the study period
Referrals to other hospital departments | 12 months of follow up from date of transplantation
  Number of referrals to other hospital departments within the study period
Referrals to general practitioner | 12 months of follow up from date of transplantation
  Number referrals to general practitioner within the study period
Referrals to municipality | 12 months of follow up from date of transplantation
  Number of referrals to rehabilitation in the municipality within the study period
Infections treated with antibiotics | 12 months of follow up from date of transplantation
  Number of infections treated with antibiotics within the study period
Number of telephone contacts to Dept. of Hematology | 12 months of follow up from date of transplantation
  Number of telephone contacts to Dept. of Hematology within the study period

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jarden, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark